CLINICAL TRIAL: NCT01682317
Title: Healthy Eating Patterns During a Lifestyle Intervention
Acronym: HEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTK IRB# FWA 6629
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Weight Loss
Keywords: eating frequency
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three Meal (Experimental): Participants in this condition will be instructed to limit their number of eating frequency to three meals per day.
  Interventions: Behavioral: Eating Frequency
- Grazing (Experimental): Participants in the increased eating frequency condition will be instructed to eat > 100 kcals every 2-3 hours.
  Interventions: Behavioral: Eating Frequency

INTERVENTIONS:
Behavioral: Eating Frequency — Thirty adults will be provided an 8-week standard lifestyle intervention, that includes a 1200-1500 kcal/day, < 30% energy from fat dietary prescription, and a physical activity goal of 200 minutes/week. Participants will be randomized to one of two conditions differing in EF using a prescription we have tested previously. One condition will limit the number of eating bouts/day to three (Three Meal), while the second condition will consume at least 100 kcal every 2 to 3 hours which should lead to approximately 6 eating bouts/day (Grazing).

SUMMARY:
The purpose of this study is to address the gap in knowledge regarding the relationship between eating frequency and weight loss.

DETAILED DESCRIPTION:
Little intervention research has been conducted to examine the influence of eating frequency (EF) on weight loss. It has been hypothesized an increased EF improves appetite control, assisting with better regulation of energy intake, thus decreasing body mass index. Unfortunately, outcomes have not shown greater appetite control with increased EF. Instead, trends favor a lower EF reducing energy intake thereby producing greater weight loss than a higher eating frequency. Thus, a lower eating frequency may lower energy intake via behavioral mechanisms. At thit time no research has examined the behavioral mechanisms that may mediate the relationship between a lower eating frequency and superior adherence to an energy-restricted diet.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* healthy overweight and obese men and women
* body mass index (BMI) between 27 and 45 kg/m squared

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR- Q)
* report being unable to walk for 2 blocks (1/4 mile) without stopping
* are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months
* diagnosed with type 1 or 2 diabetes
* have had bariatric surgery or are planning to have bariatric surgery in the next 4 months
* intend to move outside of the metropolitan area within the time frame of the investigation
* are pregnant, lactating, < 6 months post-partum, or plan to become pregnant during the investigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet | 0 and 8 weeks
  Diet (eating frequency, kilocalories, macronutrients)

SECONDARY OUTCOMES:
Ecological Momentary Assessment (EMA) | 0 and 8 weeks
  To evaluate the behavioral mechanisms of eating frequency, PalmPilot-based EMA will be used to collect real-time information on consumption cues.
Anthropometrics | 0 and 8 weeks
  Height (0 weeks only), weight and body mass index
Binge Eating | 0 and 8 weeks
  Assessed by the Eating Disorder Examination-Questionnaire (EDE-Q), which is a 36-item questionnaire derived from the Eating Disorders Examination interview.
Physical Activity | 0 and 8 weeks
  Self-reported physical activity will be assessed using the Paffenbarger Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States